CLINICAL TRIAL: NCT06791135
Title: Health and Life in Balance an Intervention to Improve Patient Capacity for Older People With Multimorbidity: A Pragmatic Mixed Methods Non-randomised Pilot Study
Brief Title: Health and Life in Balance an Intervention to Improve Patient Capacity for Older People With Multimorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 2021-04267.
Record Dates: First submitted 2025-01-13; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Multimorbidity
Keywords: Multimorbidity; Complex intervention; Person-centered care
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: Convergent Mixed-methods non-randomised pilot study
Masking Description: It is not possible to mask participating patients and health care providers. To avoid contamination we included one intervention and one control unit. In a potentially future RCT we aim to keep the cluster-design.
  In a potential future trial we aim mask outcome assessors, and researchers handling data analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Unit (Experimental): 23 participating patients in the intervention unit. These patients had the intervention Health and Life in Balance during 6 months. The intervention did not include the use of drugs or devices.
  Interventions: Other: Health and Life in Balance
- Control Unit (Placebo Comparator): 29 participating patients in the control unit. These patients had care as usual.
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: Health and Life in Balance — Health and Life in Balance is an intervention for patients 65 years and older, with 2 or more chronic diseases, and an increased care need. It involved for the patient to meet with a district nurse during 1-2 meetings to set up a care plan and then have scheduled follow-ups during 6 months. During the 1-2 meetings they went through ICAN discussion aid to discuss aspects of capacity and workload in the patient's life and healthcare. The district nurse and the patient's GP had improved communication during the intervention period.
  No use of drugs or devices was part of the intervention.
  Arms: Intervention Unit
Other: Care as usual — Care as usual
  Arms: Control Unit

SUMMARY:
The aim of this study was to examine if the intervention "Health and Life in Balance", was acceptable, feasible and if the intervention needed further development.

Health and Life in Balance is an intervention for patients 65 years and older, with 2 or more chronic diseases, and an increased care need. It involved for the patient to meet with a district nurse during 1-2 meetings to set up a care plan and then have scheduled follow-ups during 6 months. During the 1-2 meetings they went through ICAN discussion aid to discuss aspects of capacity and workload in the patient's life and healthcare. The district nurse and the patient's GP had improved communication during the intervention period.

Researchers will collect data from the patient's medical records, from questionnaires and from interviews with patients and health care providers.

Data will be analysed using both quantitative and qualitative methodologies and finally a mixed methods approach.

No drugs or devices are included in this study.

DETAILED DESCRIPTION:
Patients with multimorbidity, having more than one chronic disease, becomes more and more common as the world's population ages. However, primary care, often focusing on treating one disease at a time in short visits, show poor results in meeting these patients' needs. Hence, primary care needs to become more person-centered to meet patients with multimorbidity's needs.

In this study Health and Life in Balance, a complex intervention to improve relational continuity, person centeredness, and teamwork between the patient's district nurse and GP was piloted. The aim of the intervention was to improve patients with multimorbidity's capacity.

The aim of this study was to assess acceptability, feasibilty and need of further development of the intervention.

The study design was convergent mixed methods non randomised pilot study.

The research questions were:

1. What were the characteristics of patients recruited to the pilot study? (QUAN),
2. What components were delivered in the HLB intervention? (QUAN)
3. Was the HLB intervention associated with improvements in the proposed primary and secondary outcomes? (QUAN)
4. How did patients and health care providers experience HLB regarding participant selection, intervention content and impact on health? (QUAL)
5. What patients should HLB target and how should the intervention be delivered in a future trial? (MIXED)

Recruitment and setting:

In this study, 2 primary care units in Region Stockholm, Sweden were recruited. One was an intervention unit and the other a control unit. In both units patients 65 years and older with 2 or more chronic diseases and an increased care need were recruited by their GPs.

Intervention:

The intervention was conducted during 6 months and involved:

* Improved teamwork between the patient's GP and district nurse
* 1-2 visits with a district nurse. During the visit they went through the discussion aid ICAN. The discussion aid aims to assess patient capacity and workload from life and from health care contacts. And morst important Then they set up a care plan.
* Then they had individualised number and types of follow up contacts.

Patients in the intervention unit received the intervention and patients in the control unit received care as usual.

No drugs or devices are included in this study.

Data collection:

Quantitative data was collected in both units regarding:

1. Baseline data including age, sex, and number and types of diagnoses and medications were collected from patient medical records
2. In questionnaires by a research nurse in both units before and after the intervention. The questionnaires were:

   * Illness intrusiveness: Illness Intrusiveness Rating Scale (IIRS)
   * Treatment burden: Multimorbidity Treatment Burden Questionnaire (MTBQ)
   * Quality of Life: EuroQol -5 Dimensions- 5L (EQ-5D-5L)
   * Depressive symptoms: The Patient Health Questionnaire (PHQ-9)
   * Worry: The Penn State Worry Questionnaire (PSWQ)
   * General health: WHO Disability Assessment Schedule (WHODAS 2.0)
   * Alcohol consumption : The Alcohol Use Disorders Identification Test (AUDIT)
   * Drug consumption The Drug Use Disorders Identification Test (DUDIT)
3. Clinical outcomes was collected from patients' medical records before, and after the intervention

   * Number of medications
4. Clinical outcomes was collected from participants' medical records after the intervention was finished regarding

   * Number of visits in primary care (apart from the intervention) during the intervention period.
   * Number of visits in secondary care during the intervention period.
   * Number of admissions to hospitals during the intervention period.

Quantitative data was collected from patient medical records in the intervention unit after the intervention was finished regarding:

* Number and types of visits (part of the intervention) during the intervention
* A written care plan
* A written description of GP and DN teamwork.

Qualitative data was collected from:

* Individual interviews with participating patients in the intervention unit
* Focus group interviews with district nurses in the middle and after the intervention period.
* Focus group interviews with GPs after the intervention concluded.
* Patient medical records in the intervention unit.

Data analysis:

Quantitative data analysis:

* Descriptive statistical analyses were used to assess baseline differences between both units.
* Statistical analyses were used to assess between group differences between intervention and control group after 6 months regarding questionnaires and number of medications.

Qualitative data analysis:

* Thematic analysis by Braun and Clark was used to qualitatively analyse all qualitative data.

Mixed methods data analysis:

Quantitative and qualitative data analyses were merged together to answer the mixed methods question using joint display on interpretation level.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* 2 or more chronic diseases
* Increased care need defined by patient's GP

Exclusion Criteria:

* home health care,
* on-going treatment in a secondary unit making them unable to assimilate the intervention, for example ongoing oncological treatment,
* cognitive impairment that restricted ability to give informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Illness Intrusivenss Rating Scale | From enrollment to the end of the treatment at 6 months.
  13 items scored 1 - 7 to a total of 13 (not very intrusive) to 91 (very intrusive)

SECONDARY OUTCOMES:
Multimorbidty Treatment Burden Questionnaire | From enrollment to the end of the treatment at 6 months.
  10 items scored to a total of 0 (no burden) to 100 (>22 high burden)
EQ-5D-5L - EuroQol -5 Dimensions- 5L | From enrollment to the end of the treatment at 6 months.
  A five-dimension index score with weights derived from the English population, total -0.59 to 1, (1 representing optimal health)
PHQ-9 - The Patient Health Questionnaire | From enrollment to the end of the treatment at 6 months.
  9-items scored 0 to 3 to a total where <5 indicates absence of depressive disorder and ≥15 major depression
PSWQ - The Penn State Worry Questionnaire | From enrollment to the end of the treatment at 6 months.
  16 items scored 1 to 5, 16 is the minimal level of worry and 80 the maximum
WHODAS 2.0 - WHO Disability Assessment Schedule | From enrollment to the end of the treatment at 6 months.
  12 items scored 0 to 4, 0 points represents optimal health and 48 worst health
AUDIT - The Alcohol Use Disorders Identification Test, 12-item version | From enrollment to the end of the treatment at 6 months.
  12 items scored 0 - 5 with a total ≤ 7 suggests low-risk; 8 - 14 hazardous; ≥ 15 alcohol dependence
DUDIT - The Drug Use Disorders Identification Test | From enrollment to the end of the treatment at 6 months.
  11 items scored 0 to 4, a total score ≥25 suggests dependence
Number of medications | From enrollment to the end of the treatment at 6 months.
  Medication count from electronic list
Number of visits in primary care (apart from the intervention) | Collected post-intervention (up to 1 year)
  Visit count from medical records
Number of admissions to hospitals | Collected post-intervention (up to 1 year)
  Admission count from medical records

OTHER OUTCOMES:
Descriptive outcome - Number and types of follow-up visits | Collected post-intervention (up to 1 year)
  Number (n) of follow-up visits in A. the primary care unit B. In the patient's home C. By telephone during the intervention at the intervention unit.
  The outcome was collected from intervention participants' medical records.
Descriptive outcome - proportion of first visit(s) involving a follow-up booking | Collected post-intervention (up to 1 year)
  Proportion of 1-2 first visit (s) that involved follow-up booking. Data was collected from intervention participant's medical records.
Descriptive outcome - Number of first visit (s) | Collected post-intervention (up to 1 year)
  Number (n) of first 1-2 visits ( 1 or 2). The outcome was collected from intervention participants' medical records.
Descriptive outcome - proportion of first visit(s) involving a written care plan | Collected post-intervention (up to 1 year)
  Proportion of 1-2 first visit (s) that involved a written care plan. Data was collected from intervention participant's medical records.
Descriptive outcome - ICAN used at the initial visit(s) | Collected post-intervention (up to 1 year)
  Was ICAN filled out a the first visit(s) yes or no. The outcome was collected from intervention participants' medical records.
Descriptive outcome - Final visit offered and completed | Collected post-intervention (up to 1 year)
  Was a final visit offered and completed, yes or no. The outcome was collected from intervention participants' medical records.
Descriptive outcome - Documented GP and DN teamwork | Collected post-intervention (up to 1 year)
  Number (n) of documented communication between DN and GP about intervention participants in the intervention unit during the intervention period. Data was collected from the intervention patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Wachtler, MD, PhD, Assistant Professor, Principal Investigator — Karolinska Institute and Region Stockholm
Locations (1):
- Boo Vårdcentral, Saltsjö-Boo, Nacka, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IPD collected throughout the trial will be shared in a publication